CLINICAL TRIAL: NCT01756924
Title: Safety and Efficacy of CEM-102 With Rifampin Compared to Standard Therapy in Patients With Prosthetic Joint Infections or Spacer Infection
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: This study has been terminated; alternative study designs are being considered. Fusidic acid remains available under an Expanded Access Protocol.
Sponsor: Arrevus Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CE06-200
Record Dates: First submitted 2012-12-18; First posted 2012-12-28 (Estimated); Last update posted 2019-04-19 (Actual); Status verified 2019-04

CONDITIONS: Prosthetic Joint Infections of Hip; Prosthetic Joint Infections of Knee; Infected Spacers
Keywords: prosthetic joint infection; hip arthroplasty; MRSA; knee arthroplasty
MeSH Terms: interventions — Fusidic Acid; Vancomycin; Daptomycin; Linezolid; Rifampin; Ceftriaxone; Cefazolin; Ceftaroline; Nafcillin; Oxacillin; Ciprofloxacin; Levofloxacin; Trimethoprim, Sulfamethoxazole Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CEM-102 plus Rifampin (Experimental)
  Interventions: Drug: CEM-102; Drug: Rifampin
- Standard of Care (Active Comparator)
  Interventions: Drug: IV or Oral standard of care antibiotics

INTERVENTIONS:
Drug: CEM-102
  Other Names: fusidic acid
  Arms: CEM-102 plus Rifampin
Drug: IV or Oral standard of care antibiotics
  Other Names: vancomycin; daptomycin; linezolid; rifampin; ceftriaxone; cefazolin; ceftaroline; nafcillin; oxacillin; ciprofloxacin; levofloxacin; co-trimoxazole
  Arms: Standard of Care
Drug: Rifampin
  Arms: CEM-102 plus Rifampin

SUMMARY:
To determine if oral antibiotic treatment with CEM-102 and Rifampin is as effective and safe as the standard of care antibiotic therapy for the treatment of hip and knee prosthetic joint or spacer infections

ELIGIBILITY:
Inclusion Criteria:

* Prosthetic knee or hip joint infection
* Infected joint spacer
* Able to swallow tablets
* Able to voluntarily sign the informed consent form
* Females of childbearing potential must use an acceptable method of birth control
* The joint infection must be attributed to bacterial pathogens sensitive to fusidic acid and rifampin

Exclusion Criteria:

* History of hypersensitivity or intolerability to sodium fusidate (Fucidin®), or to rifampin
* Females who are pregnant or lactating
* Requirement for significant immunosuppression
* Bacteremia
* Known cirrhosis or decompensated liver disease
* Current treatment for HIV or Hepatitis C
* Seizure disorder, requiring anti-convulsants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2012-12; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Bacterial eradication of joint infection | 3 to 6 months
  Clinical success is defined as the absence of persistent infection in a patient who did not receive alternative antibiotic therapy targeting the infection.

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - Sarasota, Florida
  - Tamarac, Florida
  - Savannah, Georgia
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Syracuse, New York
  - Durham, North Carolina
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Charleston, South Carolina
  - Houston, Texas

REFERENCES:
- [Derived] Pushkin R, Iglesias-Ussel MD, Keedy K, MacLauchlin C, Mould DR, Berkowitz R, Kreuzer S, Darouiche R, Oldach D, Fernandes P. A Randomized Study Evaluating Oral Fusidic Acid (CEM-102) in Combination With Oral Rifampin Compared With Standard-of-Care Antibiotics for Treatment of Prosthetic Joint Infections: A Newly Identified Drug-Drug Interaction. Clin Infect Dis. 2016 Dec 15;63(12):1599-1604. doi: 10.1093/cid/ciw665. Epub 2016 Sep 28. PMID 27682068